CLINICAL TRIAL: NCT00417313
Title: Osteopuncture for Osteoarthritis-Associated Knee Pain & Disability
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AG0073; 5R21AG024288-02 (NIH)
Record Dates: First submitted 2006-12-28; First posted 2007-01-01 (Estimated); Last update posted 2007-01-01 (Estimated); Status verified 2006-12

CONDITIONS: Osteoarthritis
Keywords: knee pain; acupuncture /acupressure; alternative medicine; analgesia; arthritis therapy; chronic pain; functional ability
MeSH Terms: conditions — Osteoarthritis; Agnosia; Chronic Pain

INTERVENTIONS:
Device: periosteal electro-acupuncture (osteopuncture).

SUMMARY:
The purpose of this study is to investigate the feasibility, effectiveness, and duration of treatment response of periosteal electro-acupuncture (osteopuncture) for osteoarthritis (OA)-associated chronic knee pain.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is painful in 6.8% of men and 11.4% of women age 63-93, with over 20 million Americans affected nationwide, and may lead to a variety of untoward consequences including limitations in physical function, postural instability, sleep disturbance, psychosocial disability, and substantial utilization of health care resources. While oral analgesics represent the mainstay of treatment for chronic pain associated with knee OA, non-responders with limiting comorbidities may have few therapeutic alternatives.

The aims of this research study are to (1) reduce pain severity and disability in community-dwelling older adults with OA-associated chronic knee pain using periosteal electroacupuncture (osteopuncture), and (2) improve the physical performance, psychosocial function, sleep, and appetite of these individuals. 88 older adults with persistent knee pain and x-ray evidence of OA, no other rheumatologic disorders, no history of knee surgery, and no prominent pain in sites other than the knee(s) will be randomized to receive either osteopuncture or control osteopuncture once a week for 6 weeks. All outcome measures for pain and disability, as well as physical performance, psychosocial function, sleep, and appetite, will be collected pre-treatment, at the completion of the 6-week protocol, and 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic evidence of knee OA on a standing AP X-ray
* Bilateral knee pain for at least 3 months with pain of at least moderate intensity every day or almost every day

Exclusion Criteria:

* Non-ambulatory, or severely impaired mobility (i.e., require the use of a walker)
* Folstein Mini-Mental State Examination score of less than 24
* Severe visual or hearing impairment
* Knee pain due to factors other than OA, e.g. rheumatoid or psoriatic arthritis, gout, pseudogout, metastatic cancer
* Significant pain in parts of the body other than the knee or acute knee pain
* A large knee effusion or severe mechanical instability of the knee
* History of corticosteroid injection in the affected knee(s) during the preceding 3 months
* History of hyaluronic acid injection in the affected knee(s) during the preceding 3 months
* Acute or terminal illness
* Immune suppression
* Anticoagulation therapy
* Presence of a pacemaker
* Prior acupuncture treatment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 88
Dates: Start 2004-10; Study Completion 2006-08

PRIMARY OUTCOMES:
changes in pain and disability, measured with the Western Ontario and McMaster Universities Osteoarthritis Index

SECONDARY OUTCOMES:
changes in physical performance
psychosocial function (mood, self-efficacy, coping, fear, self-rated health)
sleep and appetite

CONTACTS AND LOCATIONS:
Overall Officials: Debra K Weiner, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Pain Evaluattion and Treatment Institute, Research Department, Pittsburgh, Pennsylvania, United States